CLINICAL TRIAL: NCT01793857
Title: Healthcare Seeking Behaviour of Primary Caregivers for Acute Otitis Media in Children Aged 6 Months to Less Than 30 Months in Panama
Brief Title: Healthcare Seeking Behaviour of Primary Caregivers for Acute Otitis Media (AOM) in Children Aged 6 Months to Less Than 30 Months in Panama
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116895
Record Dates: First submitted 2013-02-14; First posted 2013-02-18 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-09

CONDITIONS: Infections, Streptococcal
Keywords: Primary caregiver; Survey; Acute Otitis Media; Ear infection; Panama; Healthcare seeking behaviour
MeSH Terms: conditions — Streptococcal Infections; Otitis Media; Otitis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Study Group: Approximately 1300 primary caregivers of at least one child aged 6 months to less than 30 months who were interviewed during a clinic visit in Panama.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Paper questionnaire

SUMMARY:
The study is a survey aiming to describe the healthcare seeking behaviour of primary caregivers when their child aged 6 months to less than 30 months was suspected to have an episode of acute otitis media in Panama.

DETAILED DESCRIPTION:
The study is a cross sectional survey in which primary caregivers will be asked if they recall having observed an ear infection in the child in the age range 6 months to less than 30 months in the last 6 months. During the interview, the primary caregivers will be asked what they did for the child during that episode and whether they sought medical care or not. They will be also asked about the demographic characteristics (such as age range) of the child who experienced that episode and the household environment of the child at the time of the episode (such as number of household members), etc.

No questions will be asked about the episode itself if the primary caregiver does not recall that the child had one in the last six months.

Approximately 1300 primary caregivers will be interviewed in multiple clinics / well-baby clinics in Panama.

The clinics will be stratified into 'former clinical trial sites' and 'non-clinical trial sites' in urban areas of Panama, based on participation in the COMPAS trial. Both 'former clinical trial sites' and 'non-clinical trial sites' will include private and public facilities. Sites will be selected by convenience sampling and eligible subjects will be enrolled on an on-going basis, in proportion to the population coverage of each site. The participating sites have thus been stratified to be able to assess whether the healthcare seeking behaviour of primary caregivers enrolled at former clinical trial sites are different from those enrolled at non clinical trial sites.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator/interviewer believes can and will comply with the requirements of the protocol (e.g. availability of time for completion of the interview).
* Signed informed consent obtained from the subject.
* Subjects aged 18 years or above, being the primary caregiver of at least one child aged 6 months to less than 30 months, visiting a clinic.

Note:

i. Although the child will most likely be present at the time of interview, his/her presence is not required.

ii. If more than one primary caregiver fulfilling the inclusion criteria is present per child, only one will be enrolled in this study.

Exclusion Criteria:

• Subjects having previously participated in this survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary caregivers with at least one child aged 6 months to less than 30 months visiting a clinic in Panama primarily for well-baby visits or sickness visit.
Sampling Method: Non-Probability Sample
Enrollment: 1330 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Healthcare seeking behaviour of primary caregivers when their child was suspected of having an AOM episode. | During last six months before date of interview.

SECONDARY OUTCOMES:
Occurrence of suspected AOM based on symptoms reported by the primary caregiver. | During last six months before date of interview.
Potential determinants (such as access to healthcare facilities) influencing healthcare seeking behaviour of primary caregivers who suspected their child aged 6 months to < 30 months of having an AOM episode during the last six months. | During last six months before date of interview.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- Panama (13):
  - GSK Investigational Site, La Chorrera, Provincia de Panamá
  - GSK Investigational Site, Panama City, Provincia de Panamá
  - GSK Investigational Site, Arraiján
  - GSK Investigational Site, Barrio Colón
  - GSK Investigational Site, Calidonia
  - GSK Investigational Site, Curundú
  - GSK Investigational Site, El Espino
  - GSK Investigational Site, Guadalupe, La Chorrera
  - GSK Investigational Site, Juán Diaz
  - GSK Investigational Site, La Chorrera
  - GSK Investigational Site, Nuevo Arraiján
  - GSK Investigational Site, Panama City
  - GSK Investigational Site, Pueblo Nuevo